CLINICAL TRIAL: NCT01851772
Title: Feasibility Study of the Xoft® Axxent® Electronic Brachytherapy System for the Treatment of Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xoft, Inc. (Industry)
Collaborators: Icad, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRP-0010
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2015-11

CONDITIONS: Cervical Cancer
Keywords: cervical; cancer; brachytherapy; electronic; device; applicator; toxicity; gynecologic; high-dose-rate (HDR); x-ray; safety; external beam radiation therapy (EBRT)
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — Therapeutics; Brachytherapy; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects enrolled will undergo brachytherapy treatment in combination with EBRT. The maximum length of treatment will be 56 days. The treating physician will determine the appropriate course of treatment based on the physician's current practice or experience using Iridium-192 or Cesium HDR after-loaders to administer cervical brachytherapy treatments.
  Subjects enrolled will be treated with approximately 80-90 Gy total treatment dose over 4-6 fractions. Examples of commonly used dose regimens in the US are listed in section 7.6.7. This study will include data collection from the initiation of EBRT through administration of the final Xoft Axxent treatment fraction, and at one (1) month and three (3) months.
  Interventions: Device: Treatment with Electronic Brachytherapy

INTERVENTIONS:
Device: Treatment with Electronic Brachytherapy
  Other Names: Xoft®; Axxent®; Electronic; Brachytherapy; System

SUMMARY:
The purpose of this study is to evaluate the safety, performance and usability of the Xoft Axxent Electronic Brachytherapy System and Cervical Applicator as incorporated into the physician's current standard treatment practice and in replacement of high-dose-rate after-loaders using Iridium-192 or low-dose-rate Cesium treatments. Data will be collected on treatment delivery, safety, and acute toxicity.

Our hypothesis is that the treatment is safe as incorporated into the physician's current standard of practice.

ELIGIBILITY:
INCLUSION CRITERIA:

* Brachytherapy is indicated after EBRT for all cases of locally advanced disease (Stages Ib2 - IVA)
* Inoperable Stage Ia1 and Stage Ia2 may be treated with tandem-based brachytherapy alone
* Inoperable Stage Ib1 should be treated radically with brachytherapy in conjunction with EBRT. Concurrent chemotherapy may be considered at the physician's discretion and based on the presence of high risk features.
* Subjects can be treated with brachytherapy regardless of lymph node status, grade, and presence of lymphovascular invasion, tumor size, age, or histology.
* Medically fit for general or spinal anesthesia, or conscious sedation, for the insertion process
* Subjects of childbearing potential must have a negative serum pregnancy test at Screening inclusion Criteria:

EXCLUSION CRITERIA:

* Medical Contraindications to Brachytherapy (scleroderma, collagen vascular disease, active lupus )
* Prior pelvic radiotherapy with brachytherapy
* Hemoglobin level at screening < 8
* Life expectancy < 6 months

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lowndes Harrison, MD, Principal Investigator — Gadsden Regional Cancer Center
Locations (1):
- Oklahoma University, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Subjects were treated with 80-90 Gy total treatment dose over 4-6 fractions.
Period: Overall Study
Arm/Group | Treatment
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 45.67 [34 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety - Adverse Event Rate and Severity
Description: Adverse event rate and severity during and following the administration of brachytherapy treatment, through discharge from the treatment facility, and for 3 months after treatment.
Time Frame: Study Exit (90 days)
Population: Diagnosis of locally advanced cervical cancer (Stages Ib2-IVA).
Measure: Number; unit: percentage of participants and severity
Arm/Group | Treatment
Number analyzed (Participants) | 3
percentage of participants and severity
  diarrhea-mild | 100
  fatigue-mild | 100
  hot flashes-moderate | 100
  urinary track infection-mild | 33.3
  vaginal bleeding-mild | 33.3
  decreased neutrophils-mild | 33.3
  insomnia-mild | 33.3
  loss of appetite-mild | 33.3
  extremity weakness-mild | 33.3
  mucositis-mild | 33.3
  urinary frequency-mild | 33.3
  weight loss-mild | 33.3
  headache-moderate | 33.3
  chest pressure-moderate | 33.3
  light headed-moderate | 33.3
  mild skin erythema-mild | 33.3
  occasional burning with urination-mild | 33.3

2. Secondary Outcome: Device Performance
Description: Number of subjects who received complete delivery of the brachytherapy treatment using the Xoft Electronic Brachytherapy System with the cervical applicator.
Time Frame: Study Exit (90 days)
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 3
participants | 3

3. Other Pre Specified Outcome: Frequency of Adverse Events in Participants (i.e.Safety)
Description: To assess occurrence rate of radiation toxicities through three (3) months of follow-up.
Time Frame: 3 months post-Study Exit
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 3
participants | 3

ADVERSE EVENTS:
Time Frame: The type, number and severity of Adverse Events from the time of cervical brachytherapy treatment through three months follow-up.
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 3 (3)
Hoareseness (General disorders) | 1 (1)
Hot Flashes (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1) — Urinary Tract Infection
Vaginal Bleeding (Reproductive system and breast disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
Mucositis (Infections and infestations) | 1 (1)
Chest Pressure (Cardiac disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less